CLINICAL TRIAL: NCT04959409
Title: Topical Analgesia Before Inhalational Anaesthesia: A Retrospective Observational Study
Brief Title: Topical Analgesia Before Inhalational Anaesthesia
Status: Completed | Type: Observational
Sponsor: Nottingham University Hospitals NHS Trust (Other)
Responsible Party: Sponsor
Other Study IDs: 20AN008
Record Dates: First submitted 2021-06-07; First posted 2021-07-13 (Actual); Last update posted 2021-07-13 (Actual); Status verified 2021-07

CONDITIONS: Anesthesia; Pediatric ALL
Keywords: Topical analgesia; Inhalational anaesthesia
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Analgesia; Lidocaine, Prilocaine Drug Combination; Tetracaine

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Exposed Cohort: Children receiving topical analgesia
  Interventions: Drug: Topical analgesia (EMLA or AMETOP)
- Control / Unexposed Cohort: Children who do not receive topical analgesia

INTERVENTIONS:
Drug: Topical analgesia (EMLA or AMETOP) — Whether topical analgesia has or has not been administered to each child prior to them receiving an inhalational induction of anaesthesia
  Groups: Exposed Cohort

SUMMARY:
Peripheral venous cannulation (insertion of a drip line into a vein) is a fundamental component of anaesthesia for both children and adults alike. Discomfort caused by needle insertion is a common worry for children but one simple intervention that may be delivered prior to a needle insertion procedure, is the application of topical analgesia (numbing skin cream). Several creams are now available and have been found to be effective in several trials of awake children. Yet the value of these creams for children receiving an inhalational induction of anaesthesia (gas to go off to sleep before needle insertion) remains uncertain.

The aims of this study are to determine whether cream application prior to receiving gas to go off to sleep has any beneficial effects (outcomes) for children, including reduction of movement, improved needle success rates and reduced time required for needle insertion procedures. How frequently skin effects after application of the creams occur (swelling, redness, itchiness) will also be assessed.

This study will be performed as a retrospective observational study (a study which looks back in time, identifies groups of exposed (cream applied) or non-exposed (no cream applied) children and follows them over a period of time to see how their exposures affect their outcomes). Using a total population (purposive) sampling technique, 500 children from 1 month to 18 years of age undergoing elective (planned) or urgent (emergency) inhalational induction of anaesthesia (gas to go off to sleep) at Nottingham University Hospitals NHS Trust over a six month study period (August 2020 to January 2021) will be incorporated into a completely anonymised research dataset and analysed to determine whether topical analgesia (skin numbing cream) application prior to inhalational induction (gas to go off to sleep) may offer any beneficial effects for paediatric patients.

DETAILED DESCRIPTION:
This study will be performed as a retrospective cohort observational study (a study which looks back in time, identifies cohorts (groups) of 'exposed' (those who received topical analgesia (skin numbing cream)) and 'non-exposed' (those who did not receive topical analgesia (skin numbing cream)) children and follows them over a period of time to see how their exposures affect their outcomes).

Since no studies have been conducted to date, to determine the value of topical analgesia (skin numbing cream) for children receiving an inhalational induction of anaesthesia (gas to go off to sleep), this has been designed as a non-randomised preparatory study. Being non-experimental in nature, this study will attempt to evaluate preliminary null hypotheses of association. Where association(s) and/or potential benefit(s) are observed to a statistically significant level, the value and feasibility of a future experimental study, in the form of a prospective randomised controlled trial, will be evaluated.

Through acting as a first step in exploring a novel intervention, this approach is felt to offer a safe and cost-effective indication of the value a future large-scale experimental trial, which in an uninvestigated field and with only a suggestible potential for benefit, would face numerous approval challenges.

ELIGIBILITY:
Inclusion Criteria:

• All children from 1 month to 18 years of age undergoing elective or urgent inhalational induction of anaesthesia at Nottingham University Hospitals NHS Trust over a six month study period (August 2020 to January 2021)

Exclusion Criteria:

* Children receiving an attempted awake venous cannula insertion
* Children receiving an a failed intravenous induction of anaesthesia prior to an inhalational induction of anaesthesia
* Child or family history of malignant hyperthermia
* Congenital or idiopathic methaemoglobinaemia
* Glucose-6-phosphate dehydrogenase deficiency (G6PD)
* Known sensitivity to topical analgesia
* Use of analgesics within the preceding 24 hours

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: Of the children who may become study participants (identified as being eligible and not meeting the study exclusion criteria) a random sampling technique will be utilised to recruit 500 children
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-01-31 (Actual); Study Completion 2021-01-31 (Actual)

PRIMARY OUTCOMES:
Patient movement | Prospective recording by anaesthetist / member of usual care team within 30 minutes of induction of anaesthesia (with completed records stored in RCoA Logbook and Anaesthetic charts)
  To be used as a surrogate marker of pain. Movement will be defined as reflex hand and/or arm withdrawal and/or the initiation of excitatory movement(s) at the time of needle insertion

SECONDARY OUTCOMES:
FTSI (first time successful insertion) of cannula | Prospective recording by anaesthetist / member of usual care team within 60 minutes of induction of anaesthesia (with completed records stored in RCoA Logbook and Perioperative Care Record)
  Rate of FTSI (first time successful insertion) of cannula (with success defined as skin breached only once and the ability to freely instil 5 ml of normal saline intravenously (into the vein))
Overall anaesthetic time | Prospective recording by member of usual care team within 30 minutes of induction of anaesthesia (with Theatre records retrospectively analysed by research team for 'Anaesthetic Start time to (arrival in) Theatre')
  Proxy marker of duration of time to complete cannulation procedure

CONTACTS AND LOCATIONS:
Overall Officials: M Billingham, MB.ChB, Principal Investigator — Nottingham University Hospitals NHS Trust
Locations (1):
- Nottingham University Hospitals NHS Trust, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No individual participant data will be disclosed

REFERENCES:
- [Background] McMurtry CM, Pillai Riddell R, Taddio A, Racine N, Asmundson GJ, Noel M, Chambers CT, Shah V; HELPinKids&Adults Team. Far From "Just a Poke": Common Painful Needle Procedures and the Development of Needle Fear. Clin J Pain. 2015 Oct;31(10 Suppl):S3-11. doi: 10.1097/AJP.0000000000000272. PMID 26352920
- [Background] Hart D, Bossert E. Self-reported fears of hospitalized school-age children. J Pediatr Nurs. 1994 Apr;9(2):83-90. PMID 8027944
- [Background] Kortesluoma RL, Nikkonen M. 'I had this horrible pain': the sources and causes of pain experiences in 4- to 11-year-old hospitalized children. J Child Health Care. 2004 Sep;8(3):210-31. doi: 10.1177/1367493504045822. PMID 15358886
- [Background] Lee GY, Yamada J, Kyololo O, Shorkey A, Stevens B. Pediatric clinical practice guidelines for acute procedural pain: a systematic review. Pediatrics. 2014 Mar;133(3):500-15. doi: 10.1542/peds.2013-2744. Epub 2014 Feb 2. PMID 24488733
- [Background] Eccleston C, Fisher E, Howard RF, Slater R, Forgeron P, Palermo TM, Birnie KA, Anderson BJ, Chambers CT, Crombez G, Ljungman G, Jordan I, Jordan Z, Roberts C, Schechter N, Sieberg CB, Tibboel D, Walker SM, Wilkinson D, Wood C. Delivering transformative action in paediatric pain: a Lancet Child & Adolescent Health Commission. Lancet Child Adolesc Health. 2021 Jan;5(1):47-87. doi: 10.1016/S2352-4642(20)30277-7. Epub 2020 Oct 13. No abstract available. PMID 33064998
- [Background] Lander J, Hodgins M, Nazarali S, McTavish J, Ouellette J, Friesen E. Determinants of success and failure of EMLA. Pain. 1996 Jan;64(1):89-97. doi: 10.1016/0304-3959(95)00100-X. PMID 8867250
- [Background] Lander JA, Weltman BJ, So SS. EMLA and amethocaine for reduction of children's pain associated with needle insertion. Cochrane Database Syst Rev. 2006 Jul 19;(3):CD004236. doi: 10.1002/14651858.CD004236.pub2. PMID 16856039
- [Background] Manner T, Kanto J, Iisalo E, Lindberg R, Viinamaki O, Scheinin M. Reduction of pain at venous cannulation in children with a eutectic mixture of lidocaine and prilocaine (EMLA cream): comparison with placebo cream and no local premedication. Acta Anaesthesiol Scand. 1987 Nov;31(8):735-9. doi: 10.1111/j.1399-6576.1987.tb02655.x. PMID 3434165
- [Background] Maunuksela EL, Korpela R. Double-blind evaluation of a lignocaine-prilocaine cream (EMLA) in children. Effect on the pain associated with venous cannulation. Br J Anaesth. 1986 Nov;58(11):1242-5. doi: 10.1093/bja/58.11.1242. PMID 3535860
- [Background] Woolfson AD, McCafferty DF, Boston V. Clinical experiences with a novel percutaneous amethocaine preparation: prevention of pain due to venepuncture in children. Br J Clin Pharmacol. 1990 Aug;30(2):273-9. doi: 10.1111/j.1365-2125.1990.tb03775.x. PMID 2206789
- [Background] Tracey I, Mantyh PW. The cerebral signature for pain perception and its modulation. Neuron. 2007 Aug 2;55(3):377-91. doi: 10.1016/j.neuron.2007.07.012. PMID 17678852
- [Background] Otto KA. EEG power spectrum analysis for monitoring depth of anaesthesia during experimental surgery. Lab Anim. 2008 Jan;42(1):45-61. doi: 10.1258/la.2007.006025. PMID 18348766
- [Background] Otto KA, Mally P. Noxious stimulation during orthopaedic surgery results in EEG 'arousal' or 'paradoxical arousal' reaction in isoflurane-anaesthetised sheep. Res Vet Sci. 2003 Oct;75(2):103-12. doi: 10.1016/s0034-5288(03)00077-8. PMID 12893158
- [Background] Bischoff P, Kochs E, Haferkorn D, Schulte am Esch J. Intraoperative EEG changes in relation to the surgical procedure during isoflurane-nitrous oxide anesthesia: hysterectomy versus mastectomy. J Clin Anesth. 1996 Feb;8(1):36-43. doi: 10.1016/0952-8180(95)00170-0. PMID 8695077
- [Background] Hagihira S, Takashina M, Mori T, Ueyama H, Mashimo T. Electroencephalographic bicoherence is sensitive to noxious stimuli during isoflurane or sevoflurane anesthesia. Anesthesiology. 2004 Apr;100(4):818-25. doi: 10.1097/00000542-200404000-00011. PMID 15087616
- [Background] Kochs E, Bischoff P, Pichlmeier U, Schulte am Esch J. Surgical stimulation induces changes in brain electrical activity during isoflurane/nitrous oxide anesthesia. A topographic electroencephalographic analysis. Anesthesiology. 1994 May;80(5):1026-34. doi: 10.1097/00000542-199405000-00012. PMID 8017642
- [Background] Morimoto Y, Matsumoto A, Koizumi Y, Gohara T, Sakabe T, Hagihira S. Changes in the bispectral index during intraabdominal irrigation in patients anesthetized with nitrous oxide and sevoflurane. Anesth Analg. 2005 May;100(5):1370-1374. doi: 10.1213/01.ANE.0000148124.02288.D1. PMID 15845688
- [Background] Sleigh JW, Leslie K, Voss L. The effect of skin incision on the electroencephalogram during general anesthesia maintained with propofol or desflurane. J Clin Monit Comput. 2010 Aug;24(4):307-18. doi: 10.1007/s10877-010-9251-3. Epub 2010 Aug 1. PMID 20680669
- [Background] Hartley C, Poorun R, Goksan S, Worley A, Boyd S, Rogers R, Ali T, Slater R. Noxious stimulation in children receiving general anaesthesia evokes an increase in delta frequency brain activity. Pain. 2014 Nov;155(11):2368-76. doi: 10.1016/j.pain.2014.09.006. Epub 2014 Sep 10. PMID 25218826
- [Background] Antognini JF, Carstens E. Isoflurane blunts electroencephalographic and thalamic-reticular formation responses to noxious stimulation in goats. Anesthesiology. 1999 Dec;91(6):1770-9. doi: 10.1097/00000542-199912000-00031. PMID 10598621
- [Background] Kox WJ, von Heymann C, Heinze J, Prichep LS, John ER, Rundshagen I. Electroencephalographic mapping during routine clinical practice: cortical arousal during tracheal intubation? Anesth Analg. 2006 Mar;102(3):825-31. doi: 10.1213/01.ane.0000197776.26307.fa. PMID 16492836

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-04-07): https://cdn.clinicaltrials.gov/large-docs/09/NCT04959409/Prot_SAP_000.pdf